CLINICAL TRIAL: NCT00377117
Title: Diabetes Screening, Risk Management, and Disease Management in a High-Risk Mental Health Population.
Brief Title: Diabetes Screening, Risk Management and Disease Management in a High-Risk Mental Health Population Part II
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Eli Lilly and Company (Industry); St. Joseph's Health Care London (Other)
Responsible Party: Sponsor
Other Study IDs: R-05-470
Record Dates: First submitted 2006-09-14; First posted 2006-09-15 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Diabetes Mellitus; Schizophrenia; Psychotic Disorders
MeSH Terms: conditions — Diabetes Mellitus; Schizophrenia; Psychotic Disorders | interventions — Therapeutics; Mass Screening

STUDY DESIGN:
Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Management
Procedure: Screening

SUMMARY:
The purpose of this study is to learn more about the relationship between serious mental illness and the detection and management of diabetes and pre-diabetic conditions. Patients who have been diagnosed with schizophrenia are at an increased risk for developing diabetes and pre-diabetic conditions such as impaired glucose tolerance and impaired fasting glucose. In addition, novel antipsychotics have also been linked to impaired glucose metabolism and increased incidence of diabetes. The medical management of these patients may be difficult ot achieve through standard family practice. The objectives of this project are to: screen a sample of this high-risk population using an Oral Glucose Tolerance Test (OGTT), and to provide multidisciplinary team support to those identified as having diabetes or a pre-diabetic condition.

DETAILED DESCRIPTION:
Many studies suggest that the extensive psychiatric needs of some patients could take attention away from management of other health problems and from the usual health promotion services physicians provide. Studies suggest that medical comorbidity has often been under recognized and under diagnosed in psychiatric patients, especially among those with schizophrenia. Unrecognized physical diseases are often associated with serious, potentially fatal illness, and may exacerbate the symptoms of psychiatric illness.

The disorder of schizophrenia has been repeatedly associated with a higher than normal incidence of medical illnesses- specifically, diabetes mellitus (DM). The prevalence of DM in a retrospective study of 95 chronic schizophrenic patients was found to be 15.8% - 4 to 5 times higher than that reported in epidemiological surveys in the general population. This increased risk has recently been formally recognized in the Canadian diabetes practice guidelines. In addition, the first line treatment of schizophrenia as per many published clinical practice algorithms, novel antipsychotics (NAP), has been associated independently with increased risk for diabetes. Novel antipsychotics such as clozapine, olanzapine, quetiapine, and risperidone have demonstrated efficacy in the treatment of schizophrenia with generally fewer extrapyramidal side effects than high dosed typical neuroleptics. However, there is accumulating data suggesting that treatment with at least some of the NAPs may be associated with the development of DM and associated risk factors. The use of olanzapine, for example, has been associated with weight gain, exacerbation of previously well-controlled diabetes, and onset of type 1 and type 2 diabetes. Clozapine has also been associated with weight gain in several reports, as well as increased risk of developing diabetes, and at least one report citing deaths from diabetic ketoacidosis after long-term use.

High-risk groups need targeted diabetes strategies. The Canadian diabetes practice guidelines outline that the service model needed to achieve the benchmarks set for diabetes care will need to be designed to reflect the unique diabetes related challenges faced by various segments of the diabetes epidemic. Diabetes care should be organized around a multidisciplinary diabetes healthcare (DHC) team that can establish and sustain a communication network between the person with DM and the necessary healthcare and community systems. The high risk mental health communities in Ontario need a targeted primary health care service delivery model that attends to the unique set of diabetes related challenges they face, including: weight increase related to medication use, inadequate self-care resources and capacity related to poverty, social constraints and lack of supports, communication barriers and mental health symptomology impacting interactions with service providers.

Current guidelines for diabetes management are clear regarding the monitoring and treatment of identified high-risk groups. Screening for DM should be performed every three years in individuals over 40 years of age. However, more frequent and/or earlier testing with a 75-g Oral Glucose Tolerance Test (OGTT) should be considered in people with identified risk factors such as schizophrenia and NAP use. Annual screening could detect individuals with undiagnosed DM as well as individuals with the pre-diabetic conditions of Impaired Fasting Glucose and Impaired Glucose Tolerance. Results of large, well-designed studies assessing early interventions in adults to prevent the progression from pre-diabetic conditions to DM have recently been published. These studies have demonstrated significant risk reduction with lifestyle management and appropriate pharmacologic interventions. It is also well documented that a comprehensive multidisciplinary Diabetes Healthcare team can help slow the progression of the disease and reduce the incidence of DM-related complications for those already diagnosed with DM.

The London Intercommunity Health Centre (LIHC) has recently piloted a diabetes program addressing the needs of a high-risk mental health population within the recommended guidelines. The program was designed as a "one stop shop" for self-management teaching, medication and glucose monitoring, and referral to specialist providers as needed. The structure of the program followed the Canadian Diabetes Association Clinical Practice Guidelines. Although the program has yet to be implemented long enough to determine if the progression from pre-diabetes to diabetes was prevented, pre-diabetic patients involved in the program have demonstrate clinically significant improvement in lipid profiles and blood pressure measurements. Those patients diagnosed with DM, who participated in the program, were found to attend regularly, and demonstrated a clinically significant improvement in their metabolic control. Thus, initial results from the LIHC, and a recent extension of this model into a community population, indicate that this model of diabetes care for this high-risk mental health population is promising for diabetes risk and disease management.

ELIGIBILITY:
Inclusion Criteria:

* Patients active in current Regional Mental Health Care London, Specialized Adult London Ambulatory Care and Assertive Community Treatment programs with known diagnosis of a Psychotic Disorder and/or use of Novel Antipsychotics.
* Must have family physician contact and ability to consent to medical care.

Exclusion Criteria:

* Any patient with declaration on file stating incapable of consenting to medical treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2006-05 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stewart B Harris, MD MPH CCFP FACPM, Principal Investigator — Centre for Studies in Family Medicine; David RS Haslam, MSc MD FRCPC, Principal Investigator — St. Joseph's Health Care London
Locations (1):
- Regional Mental Health Care London, London, Ontario, Canada

REFERENCES:
- [Background] Crews C, Batal H, Elasy T, Casper E, Mehler PS. Primary care for those with severe and persistent mental illness. West J Med. 1998 Oct;169(4):245-50. PMID 9795595
- [Background] Brown JB, Lent B, Stirling A, Takhar J, Bishop J. Caring for seriously mentally ill patients. Qualitative study of family physicians' experiences. Can Fam Physician. 2002 May;48:915-20. PMID 12053636
- [Background] Kushner K, Diamond R, Beasley JW, Mundt M, Plane MB, Robbins K. Primary care physicians' experience with mental health consultation. Psychiatr Serv. 2001 Jun;52(6):838-40. doi: 10.1176/appi.ps.52.6.838. PMID 11376238